CLINICAL TRIAL: NCT05388955
Title: A Pre-transplantation Risk Assessment Tool for Graft Survival After Pediatric Kidney Transplantation Based on 1425 Dutch Transplantations
Brief Title: Risk Assessment Tool for Graft Survival in Pediatric Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Riskcalculator.Pediatric.ntx
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2022-05

CONDITIONS: Kidney Transplant Failure and Rejection; Pediatric Kidney Disease
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None, transplantation recipients — None, observational

SUMMARY:
Registry study in which data of all pediatric kidney recipients in the Netherlands (registered in the Nederlandse Orgaan Transplantatie Registry) are studied to develop a risk calculator for graft loss.

DETAILED DESCRIPTION:
The pre-transplantation parameters of all recipients are used to do a multivariable regression analysis.

The B-coefficients of this analysis will be used to develop a risk calculator that predicts graft survival after transplantation per year of transplantation.

ELIGIBILITY:
Inclusion Criteria:

Pediatric kidney recipients

* transplantation in the Netherlands
* signed informed consent

Exclusion Criteria:

* combined transplantation (pancreas-kidney of liver-kidney transplantation)
* No informed consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric kidney recipients that received their kidney <18 years in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 1425 (Actual)
Dates: Start 1966-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Graft survival | Up to 50 years after transplantation
  Functioning graft of death with functioning graft. Survival graph: Percentage recipients with a functioning graft over time

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth De Wall, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No
Not owner of the data, NOTR owns the data

REFERENCES:
- [Derived] Oomen L, de Jong H, Bouts AHM, Keijzer-Veen MG, Cornelissen EAM, de Wall LL, Feitz WFJ, Bootsma-Robroeks CMHHT. A pre-transplantation risk assessment tool for graft survival in Dutch pediatric kidney recipients. Clin Kidney J. 2023 Mar 23;16(7):1122-1131. doi: 10.1093/ckj/sfad057. eCollection 2023 Jul. PMID 37398686